CLINICAL TRIAL: NCT01350921
Title: A Sequential, Open Label Study to Compare the Pharmacokinetics, Safety and Tolerability of Ticagrelor and Venlafaxine Given Concomitantly in Healthy Subjects Aged 18 to 45 Years
Brief Title: Evaluation of the Drug-drug Interaction Between Ticagrelor and Venlafaxine When Taken Together in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5130C00073
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Drug Drug Interaction
Keywords: phase 1; ticagrelor; venlafaxine
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ticagrelor — 90 mg oral immediate release tablets, single dose on days 1 and 9
Drug: Venlaflaxin — 37.5 mg oral immediate release tablets, administered twice daily on days 4-8

SUMMARY:
Study evaluates the drug-drug interaction between Ticagrelor and Venlafaxine when taken together in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* a weight of at least 50 kg and a body mass index between 18 to 30 kg/m2

Exclusion Criteria:

* History of clinically significant disease or disorder as judged by the investigator
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of drug.
* History of haemophilia, von Willebrand´s disease, lupus anticoagulant or other diseases/syndromes that may alter or increase bleeding.
* History of previous or ongoing psychiatric disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
area under the plasma concentration-time curve during a dosing interval (AUCτ) and observed maximum plasma concentration (Cmax) | Multiple assessments during day 8 and 9.
  Venlafaxine and O-desmethylvenlafaxine (ODV) on Day 8 (after multiple dose administration of venlafaxine for 4 days) and Day 9 (after concomitant administration of venlafaxine and ticagrelor):

SECONDARY OUTCOMES:
Venlafaxine and ODV on Days 8 and 9: time to Cmax (tmax) | Multiple assessments during day 1 and 9-11
  Ticagrelor and AR-C124910XX on Day 1 (after single dose administration of ticagrelor) and Day 9 (after concomitant administration of venlafaxine and ticagrelor): area under the plasma concentration-time curve from zero to infinity (AUC), Cmax, tmax and apparent terminal half-life t½λz
Safety and tolerability of ticagrelor and venlafaxine when given concomitantly by assessments of amount of adverse events | Multiple assessments from day -1 do day 12 and a single assessment at follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Horrow, PhD, Study Director — AstraZeneca Wilmington; Mirjana Kujacic, PhD, Study Chair — AstraZeneca Mölndal; Kelli Craven, MD, Principal Investigator — Quintiles Kansas Overland Park US
Locations (2):
- Research Site, Overland Park, Kansas, United States
- Research Site, Uppsala, Sweden